CLINICAL TRIAL: NCT03907150
Title: Interest of Strain Ultrasound in the Diagnosis of Pneumothorax: Prospective Multicenter Observational Study
Brief Title: Pleurostrain: Interest of Strain Ultrasound in the Diagnosis of Pneumothorax
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Xavier Bobbia, Principal Investigator, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: XBobbia/Pleurostrain
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Pneumothorax
Keywords: Pont-of-Care Ultrasound
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumothorax: Pneumothorax
  Interventions: Diagnostic Test: Strain ultrasound
- Normal: Normal lung
  Interventions: Diagnostic Test: Strain ultrasound

INTERVENTIONS:
Diagnostic Test: Strain ultrasound — Post-interpretation of recorded ultrasound loops

SUMMARY:
The objective of this study is to investigate whether the use of strain ultrasound can improve the lung ultrasound accuracy for the diagnosis of pneumothorax, particularly for inexperienced physicians.

DETAILED DESCRIPTION:
Prospective multi-centre diagnostic study based on the post-interpretation of recorded ultrasound loops as part of standard patient management.

ELIGIBILITY:
Inclusion Criteria:

* Age over 17 years old
* Management in an investigative centre
* Presenting a suspicion of pneumothorax
* Having had a pulmonary ultrasound scan
* Having had a CT scan within 2 hours after or before the pulmonary ultrasound

Exclusion Criteria:

* Pregnant or breastfeeding women
* Persons not covered by a social security scheme
* Persons deprived of their liberty
* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under the protection of justice, guardianship or curatorship
* Patient refuses to participate
* It is impossible to give informed information about
* The patient does not read French fluently
* Patient with any known pulmonary pathology pre-existing prior to the hospitalization episode
* Patient with a lung condition other than pneumothorax on a scanner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department or critical care patient who had a chest CT within 2 hours
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Pneumothorax diagnosis by an inexperienced physician in lung ultrasound | May 1, 2021
  The main endpoint will be a binary qualitative value: diagnosis of pneumothorax (yes/no) judged by inexperienced physicians performing pleural strain.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital La Timone, Marseille
  - AP-HM - Hopital Nord, Marseille
  - CHU Nîmes, Nîmes
  - Nimes University hospital, Nîmes